CLINICAL TRIAL: NCT04664582
Title: Sentinel Lymph Node Biopsy for Cutaneous Squamous Cell Carcinoma of the Head and Neck - A Multi-Institutional Prospective Study
Brief Title: Sentinel Lymph Node Biopsy for Cutaneous Squamous Cell Carcinoma of the Head and Neck
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sena Turkdogan, Principal Investigator, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLNB for SCC
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Sentinel Lymph Node
MeSH Terms: interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Masking Description: Treatment with sentinel lymph node biopsy cannot be masked for the participant, care provider, nor investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sentinel Lymph Node Biopsy (Experimental): Lymphoscintigraphy will be ordered alongside usual pre-operative investigations. Intra-operatively, the excision of the primary tumor will be done with the aim of histologically clear margins and appropriate closure as per routine practice at the operating surgeon's discretion. The patients are injected with technicium 99 pre-operatively and a sentinel lymph node biopsy will be performed with a handheld gamma probe.
  Interventions: Procedure: Sentinel Lymph Node Biopsy
- Standard of Care (No Intervention): These patients will be treated with standard of care, which is wide local excision of the primary tumor without performance of sentinel lymph node biopsy, if not indicated.

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — see intervention group description
  Arms: Sentinel Lymph Node Biopsy

SUMMARY:
Current guidelines in management of regional lymph node metastases for cSCC patients include surgical resection with or without adjuvant therapy as well as chemotherapy and interdisciplinary management; in advanced disease, supportive and palliative care is recommended. These guidelines also define the role of SLNB in management of high-risk cSCC as unclear and suggest further studies need to determine its utility and indications11.

Currently, routine practice of performing SLNB in cSCC varies across Quebec and within Canada. At many institutions, SLNB is not routinely performed on patients with cSCC. The current standard of treatment is to observe closely when a patient is deemed to have a high-risk cancer, and if they have clinical or radiological findings of lymphadenopathy, a formal surgical neck dissection is performed. Given the comorbidities and risks involved in treatment of regional lymph nodes in cSCC, the role of SLNB in cSCC patients needs further clarification. This multicentre prospective study aims to better clarify this role and formulate suggested criteria for its indications.

DETAILED DESCRIPTION:
INTRODUCTION:

Cutaneous Squamous Cell Carcinoma (cSCC) is a malignant neoplasm that arises from epidermal keratinocytes. It is the second most commonly seen nonmelanoma skin cancer after basal cell carcinoma (BCC) and is one of the most common malignancies in the world. The annual incidence of nonmelanoma skin cancers exceed all other malignancies combined. It also has a predilection for the head and neck, due to being a common location for sun-exposed skin. While incidences of both BCC and squamous cell carcinoma are increasing worldwide, cSCC is increasing even more disproportionately. This increase in skin cancer trends is likely due to a combination of factors including increased sun exposure along with increasing life expectancies. Furthermore, unlike BCC which tends to have an indolent course and is rarely metastatic, cSCC has more metastatic potential than BCC. While the vast majority of cSCC cases can be treated with curative intent without complication, there are a certain subset of cSCC which behave aggressively with significant risk for local recurrence and distant metastasis.

Many retrospective studies have tried to define "high-risk" features in cSCC that are predictive of regional and distant metastasis or poor survival, including local recurrence, depth of invasion, larger size, perineural and lymphovascular invasion, poor differentiation, and immunosuppression. Despite this, there is poor concordance in current guidelines on which patient and tumor characteristics constitute high-risk features. These include discrepancies between major guiding associations, such as the American Joint Committee on Cancer and National Comprehensive Cancer Network Clinical Practice Guidelines. Ultimately, a consensus on the definition of high-risk features of cSCC is necessary in order to produce practical and precise guidelines to enhance patient care.

Sentinel Lymph Node Biopsy (SLNB) is an established prognostic procedure in determining the degree of spread of malignant cells. It is used widely in skin cancers such as melanoma, with consistent recommended guidelines by the American Society of Clinical Oncology (ASCO) and Society of Surgical Oncology (SSO). However, no such guideline currently exists for cSCC and recommendations for its routine use is conflicting in the literature. There exist many studies concerning the use of SLNB in cSCC, most of which are small and retrospective in nature.

Two systematic reviews on the subject both revealed that prospective studies documenting high-risk features were necessary. A meta-analysis that included 36 studies by Thompson et al. narrowed down tumor depth and tumor diameter as having the most significant risk ratio for recurrence, metastasis, and disease-specific death in cSCC respectively. However, they also concluded that unified, consistent collection and reporting of risk factors in a prospective, multicentered effort was needed. Lastly, a multi-institutional prospective study was performed by Mooney at al between 2010-2017. While the study was well designed, they only looked at 5 tumor characteristics, including tumor site, diameter, depth, differentiation and invasion. It also appears that they used a blue dye technique for SLNB over radioactive tracer methods preferred at other institutions. They conclude that significant predictors of metastasis were four or more high-risk features, which may be vague depending on which predictors the treating team is considering. Furthermore, the generalizability of the study may be limited due to including only Australian institutions. No prospective multi-institutional studies have looked at a North American patient population.

This prospective multicentre study aims to clarify the role of SLNB in cSCC by identifying patient and tumour characteristics for candidacy criteria in SLNB indication.

RATIONALE:

After the introduction of SLNB by Morton and Cochran in the 1990s, many studies and trials were run to determine its role and indications, particularly in melanoma. Three landmark trials, MSLT-I, DeCOG-SLT and MSLT-II, among other studies, lead to the creation of SLNB guidelines by ASCO and SSO for melanoma patients. SLNB has been shown to provide substantial prognostic information as well as possible therapeutic effects in some cases; whereas Completion Lymph Node Dissection (CLND) has been demonstrated not to provide any survival benefits.

Current guidelines in management of regional lymph node metastases for cSCC patients include surgical resection with or without adjuvant therapy as well as chemotherapy and interdisciplinary management; in advanced disease, supportive and palliative care is recommended. These guidelines also define the role of SLNB in management of high-risk cSCC as unclear and suggest further studies need to determine its utility and indications.

Currently, routine practice of performing SLNB in cSCC varies across Quebec and within Canada. At many institutions, SLNB is not routinely performed on patients with cSCC. The current standard of treatment is to observe closely when a patient is deemed to have a high-risk cancer, and if they have clinical or radiological findings of lymphadenopathy, a formal surgical neck dissection is performed. Given the comorbidities and risks involved in treatment of regional lymph nodes in cSCC, the role of SLNB in cSCC patients needs further clarification. This multicentre prospective study aims to better clarify this role and formulate suggested criteria for its indications.

ELIGIBILITY:
Inclusion Criteria: high risk features rendering the patient eligible for SLNB in this study will include two or more of the following clinical or pathological features:

* Immunocompromised
* Size more than 2 cm
* Depth more than 6 mm
* Poorly differentiated histology
* Perineural invasion > 0.1mm
* Extensive lymphovascular invasion

Exclusion Criteria:

* Evidence of lymph node metastasis (clinical, radiological, or pathological)
* Previous surgery altering lymphatic drainage of the head and neck, such as a prior neck dissection or prior neck irradiation
* Pregnancy of breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
predictive value of sentinel lymph node biopsy in cutaneous squamous cell carcinoma | 1 month after feasibility recruitment completed (anticipated Dec 2021)

SECONDARY OUTCOMES:
disease free five year survival | 5 years post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mlynarek, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No